CLINICAL TRIAL: NCT00905879
Title: Observational Study on the Safety and Tolerability of Gadobutrol (Gadovist) Among Filipino Patients
Brief Title: Observational Study on the Safety and Tolerability of Gadobutrol (Gadovist) Among Filipino Patients in Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer HealthCare AG
Other Study IDs: 13926; GV0811PH (Other: Company Internal)
Record Dates: First submitted 2009-04-27; First posted 2009-05-21 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Magnetic Resonance Imaging
Keywords: Magnetic Resonance Imaging (MRI); Observational study; Gadobutrol
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Gadobutrol (Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadovist, BAY86-4875) — Patients who will need to undergo contrast enhanced MRI with gadobutrol (Gadovist)

SUMMARY:
Patients will be recruited from those who will undergo contrast enhanced MRI. Safety and tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above undergoing contrast enhanced cranial or spinal MRI with Gadobutrol (Gadovist)

Exclusion Criteria:

* History of hypersensitivity reaction to gadolinium containing contrast material
* Hypersensitivity to any of the ingredients of Gadobutrol (Gadovist)
* History of hypersensitivity to any other contrast agent
* Patients with uncorrected hypokalemia
* Pregnant and lactating women
* Patients with severe cardiovascular diseases
* Patients in whom MRI cannot be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years old and above who will undergo contrast enhanced MRI with Gadobutrol (Gadovist)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-06; Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures would be safety and tolerability of Gadovist which would be measured by change in Vital signs before and after the procedure and the occurrence of serious or non-serious adverse events | Up to 1 hour after MRI

OTHER OUTCOMES:
Magnetic field strength of MRI | During the procedure
Volume of contrast agent used | During the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Philippines